CLINICAL TRIAL: NCT04299854
Title: Modalités de Déclenchement Des Patientes Obèses à Terme (MODOBAT)
Brief Title: Modality of Induction of Labor in Obese Women at Term (MODOBAT)
Acronym: MODOBAT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/469
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-03

CONDITIONS: Induction of Labor Affected Fetus / Newborn; Obese
Keywords: Induction of Labor; BMI; Obesity; caesarean; C-section; Pregnancy; Balloon; Dinoprostone
MeSH Terms: conditions — Obesity | interventions — Dinoprostone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- Vaginal Dinoprostone: Induction of labor by 10mg of vaginal dinoprostone
  Interventions: Drug: Dinoprostone 10mg
- Single Balloon Foley Catheter: Induction of labor by single balloon Foley catheter
  Interventions: Device: single balloon Foley catheter

INTERVENTIONS:
Drug: Dinoprostone 10mg — Vaginal delivery system containing 10mg of dinoprostone placed at the bottom of the vagina
  Groups: Vaginal Dinoprostone
Device: single balloon Foley catheter — A single balloon Foley catheter is being inserted on transcervical and inflated above the internal cervical os
  Groups: Single Balloon Foley Catheter

SUMMARY:
In normal-weight patients, numerous studies show an equivalence of efficacy between dinoprostone and balloon to induce labor. In obese patients, this efficacy is not known, although inductions of labor are more frequent. MODOBAT aims to describe the ability to obtain a vaginal delivery of two modality of induction of labor (vaginal dinoprostone and single balloon Foley catheter) in obese women at term.

DETAILED DESCRIPTION:
Obesity has for several decades become a global epidemic in developed countries. In case of pregnancy, obesity leads to an increased risk of obstetric complications, the indications of induction of labor are then more frequent. Unfortunately the rate of failed induction is also higher and therefore the risk of caesarean section is increased in obese women compared to normal-weight patients when induction of labor is indicated. However, in this context effectiveness of each mode of induction is not known. Some retrospective studies would suggest that the balloon would be more effective because it would not be affected by the increase in fat mass but this result are not , but the to confirm this hypothesis.

The aim of this study is to describe the caesarean section rate in induction of labor by vaginal dinoprostone and single balloon Foley catheter in obese women. Patients in the vaginal dinoprostone arm will be included retrospectively and patients in the single balloon Foley catheter arm will be included prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Medical indication of induction of labor
* BMI ≥ 30 kg / m2
* Bishop < 6
* Singleton
* Gestational age > 36 SA + 6j
* Cephalic presentation

Exclusion Criteria:

* Adults under guardianship or curatorship
* Scarred uterus
* Placenta praevia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients of the level III maternity of university hospital center of Besançon and level IIB maternity of regional hospital of Trevenans, France.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Cesarean sections | 1 year
  Rate of cesarean sections in each group

SECONDARY OUTCOMES:
Entry into active phase (dilation to 5-6 cm) | 1 year
  Rate of entry into active phase (dilation to 5-6 cm)
Complication | 1 year
  Complication rate = composite criteria including :
  * Hypercinesia / hypertonia rate
  * Rate of fetal heart rate anomalies
  * Fever rate during work
  * Rate of uterine ruptures
  * Postpartum hemorrhage rate
  * Rate of infectious complications in immediate postpartum (fever> 38.5 ° or wall abscess or endometritis defined by a fever greater than 38 ° with pain in uterine mobilization and foul or foul-smelling lochia)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Besançon, Besançon
  - Hopital Nord Franche-Comté, Trévenans